CLINICAL TRIAL: NCT00954434
Title: Effects of Red Wine on Cardiovascular Risk Factors in Humans
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University Hospital, Linkoeping (Other)
Responsible Party: Fredrik H Nystrom MD, professor, University Hospital, Linkoeping, Sweden
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: M246-08
Record Dates: First submitted 2009-08-06; First posted 2009-08-07 (Estimated); Last update posted 2016-05-17 (Estimated); Status verified 2016-05

CONDITIONS: Healthy Subjects

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- red wine (Experimental): intervention: dietary supplement intake of red wine on a daily basis, 1 glass/day for women, 2 for men
  Interventions: Dietary Supplement: red wine
- total abstention from alcohol (No Intervention)

INTERVENTIONS:
Dietary Supplement: red wine — intake of red wine on a daily basis
  Arms: red wine

SUMMARY:
Fifty healthy human subjects are randomized to not to consume any alcohol at all or to drink 1 glass of red wine/day for women or 2 glasses for men for three months. Outcomes are changes in mood, blood lipids, insulin levels, markers of inflammation and effects on liver and body composition.

ELIGIBILITY:
Inclusion Criteria:

* healthy subjects
* 25 years of age and older

Exclusion Criteria:

* alcoholic first degree relatives

Ages: 25 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2009-09; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
effects on laboratory variables, mood and body composition | 3 months
  changes in mood, blood lipids, insulin levels, markers of inflammation and effects on liver and body composition.

SECONDARY OUTCOMES:
effects on liver fat amount | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Fredrik H Nystrom, MD PhD prof, Principal Investigator — University Hospital of Linkoping, Sweden